CLINICAL TRIAL: NCT03056183
Title: Care Transitions for Medically Ill Patients With Depression
Brief Title: Care Transitions for Patients With Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Waguih William IsHak, MD, FAPA, Vice Chair, Education and Research, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045116
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Patients in the Depression Care Transitions intervention will have a Transitional Care Social Worker who will maintain daily phone contact, home visits, and will attend with the patient medical and psychiatric appointments for an average of three months following discharge. Patients in the usual care group will proceed as usual (scheduled follow-up visits). These subjects will also be asked to complete questionnaires relating to quality of life and physical and mental health status.
  Interventions: Behavioral: Depression Care Transitions (DCT)
- Control Group - Standard of Care (No Intervention): To be followed per standard of care and data from their medical records will be reviewed.

INTERVENTIONS:
Behavioral: Depression Care Transitions (DCT) — DCT Intervention group - Patients in the DCT intervention will have a Transitional Care Social Worker (TCSW) who will maintain daily phone contact, home visits, and will attend with the patient medical and psychiatric appointments for an average of three months following discharge. Patients in the usual care group will proceed as usual (scheduled follow-up visits). These subjects will also be asked to complete questionnaires relating to quality of life and physical and mental health status.
  Arms: Treatment Group

SUMMARY:
Aim 1: To collect data on a Depression Care Transition (DCT) program's association with self-care behaviors as measured by medication adherence and clinic visit attendance, after discharge. Hypothesis 1: Compared with usual care, patients who receive the DCT intervention will have significantly greater medication adherence and clinic visit attendance, at 30, 90, and 365 days after discharge.

Aim 2: To collect data on DCT's association with clinical/health outcomes as measured by depression severity, functional status, and overall physical and mental health, after discharge. Hypothesis 2: Compared with usual care, patients who receive the DCT intervention will have significantly larger improvements in depression severity, functional status, and overall physical & mental health at 30, 90, and 365 days after discharge.

Aim 3: To collect data on DCT's association with utilization outcomes as measured by readmissions, length of subsequent hospital stays, and cost of care, after discharge. Hypothesis 3: Compared with usual care, patients who receive the DCT intervention will have significantly lower hospital readmissions, shortened length of subsequent hospital stays and lower cost of care, at 30, 90, and 365 days of discharge.

Leading the research team are a psychiatrist (Dr. IsHak - PI) and a hospitalist (Dr. Nuckols - Co-I) with an advanced and well-established track record of health services research/scholarship in the fields of depression, outcome measurement, and economic implications of improving the quality and safety of health care.

DETAILED DESCRIPTION:
This study will contribute to advancing the science of continuity of care delivery for depressed medical inpatients by collecting data on the impact of a modified evidence-based care transition model on clinical/health and utilization outcomes of depression in medically ill inpatients. The study could generate evidence to support the inpatient application of the USPSTF guidelines for screening adults for depression through staff-assisted depression care systems including follow-up and continuity of care. This study will add to the existing outpatient evidence for identification and treatment of depression in improving outcomes (Simon et al., 2001;O'Connor et al., 2013), the crucial aspect of inpatient evidence for depression identification, treatment, and continuity of care/care transitions in improving clinical/health and utilization outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than the age of 18, admitted to Cedars-Sinai Medical Center, English speaking, and answers "yes" to either question on the PHQ-2 instrument.

Exclusion Criteria:

* Participants under the age of 18, non-English speaking, and does not answer "yes" to either question on the PHQ-2 instrument.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Transitional Care | 365 days
  Patients in the DCT intervention will have a Transitional Care Social Worker (TCSW) who will maintain daily phone contact, home visits, and will attend with the patient medical and psychiatric appointments for an average of three months following discharge. Patients in the usual care group will proceed as usual (scheduled follow-up visits). These subjects will also be asked to complete questionnaires relating to quality of life and physical and mental health status.

SECONDARY OUTCOMES:
Depression Surveys | 365 days
  All patients who are admitted to CSMC are screened for depression using the PHQ instrument (Kroenke, Spitzer, & Williams, 2001). Patients are asked two questions about frequent occurrence of cardinal depressive symptoms - sadness and anhedonia - and provide yes/no answers to the intake nurse (PHQ-2). If patients answer, "yes" to either question, they are administered the complete PHQ-9 instrument. Per the CSMC depression screening protocol, if patients score >12 on the PHQ-9, a social worker evaluation, and notification of the admitting physician and psychiatry, will take place. The subjects will be identified through the psychiatrist who will discuss the risks and benefits of study participation, and assess the patient's interest in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Waguih IsHak, MD, Principal Investigator — Cedars-Sinai Medical Center

IPD SHARING:
Plan to Share IPD: No